CLINICAL TRIAL: NCT05737173
Title: Comparison Efficacy of Intraarticular Knee Injection in Knee Osteoarthritis With Leukocyte-rich and Leukocyte-poor Platelet-rich Plasma
Brief Title: Intraarticular Leukocyte-rich and Leukocyte-poor PRP for Osteoarthritis of the Knee
Acronym: PRP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 023/2563
Record Dates: First submitted 2023-02-12; First posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Osteo Arthritis Knee
Keywords: OA knee; PRP; Leukocyte concentration; Osteoarthritis Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Leukocyte-rich platelet-rich plasma (Experimental): Leukocyte-rich PRP: Centrifuge at 300 G for 5 min, separate the plasma and buffy coat layers, and then centrifuge at 700 G for 17 min with calcium chloride at the ratio of 1:5 to PRP by volume.
  Interventions: Drug: Leukocyte-poor platelet-rich plasma; Drug: Corticosteroid
- Leukocyte-poor platelet-rich plasma (Experimental): Leukocyte-poor PRP: Centrifuge at 123 G for 15 min, separate the plasma and buffy coat layers, and then centrifuge at 448 G for 10 min. Calcium chloride was added 1:5 to PRP by volume.
  Interventions: Drug: Leukocyte-rich platelet-rich plasma; Drug: Corticosteroid
- Corticosteroid (Experimental): Corticosteroid: 1 ml of triamcinolone acetonide (40mg/ml) mixed with 0.9% NaCl to a total volume of 4 ml.
  Interventions: Drug: Leukocyte-rich platelet-rich plasma; Drug: Leukocyte-poor platelet-rich plasma

INTERVENTIONS:
Drug: Leukocyte-rich platelet-rich plasma — Intra-articular knee injection
  Other Names: LRPRP
  Arms: Corticosteroid; Leukocyte-poor platelet-rich plasma
Drug: Leukocyte-poor platelet-rich plasma — Intra-articular knee injection
  Other Names: LPPRP
  Arms: Corticosteroid; Leukocyte-rich platelet-rich plasma
Drug: Corticosteroid — Intra-articular knee injection
  Other Names: CS
  Arms: Leukocyte-poor platelet-rich plasma; Leukocyte-rich platelet-rich plasma

SUMMARY:
To compare the efficacy of intraarticular knee injection between leukocyte-rich and leukocyte-poor platelet-rich plasma in knee osteoarthritis treatment

DETAILED DESCRIPTION:
Participants were randomized into 3 groups (leukocyte-rich platelet-rich plasma (LR-PRP), leukocyte-poor platelet-rich plasma (LP-PRP), and Corticosteroid (CS)). The primary outcome of this study is The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and was measured pre-treatment and post-treatment at follow-up at 1, 3, and 6 months

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years old, Plain radiographs knee AP shows Kellgren-Lawrence classification 1-4, Refuse the use of NSAIDs for 2 weeks.

Exclusion Criteria:

* 1) Previous intra-articular injection therapy in the past 6 months; 2) Previously treated with intra-knee PRP injection; 3) History of knee arthritis from other causes such as rheumatoid arthritis, pseudogout or infectious joints 4) History of blood disorder including anemia and thrombocytopenia (Hb < 12 g/dl, plt < 150,000/ml ) 5) History of surgery on the aforementioned knee 6) Obvious knee deformity (valgus > 15, varus > 20, flexion ROM < 90 , extension lag > 20) 7) Pregnancy and lactation

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 6 months
  a self-administered questionnaire consisting of 24 items divided into 3 subscales
  Pain (5 items) Stiffness (2 items) Physical Function (17 items)

SECONDARY OUTCOMES:
VAS pain | 6 months
  total of 10 score
the time up and go test | 6 months
  unit: second
30-second chair stand test | 6 months
  unit second

CONTACTS AND LOCATIONS:
Overall Officials: Surapol Athiprayul, MD, Study Director — Queen Savang Vadhana Memorial Hospital, Thailand
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Si Racha, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kuptniratsaikul V, Tosayanonda O, Nilganuwong S, Thamalikitkul V. The epidemiology of osteoarthritis of the knee in elderly patients living an urban area of Bangkok. J Med Assoc Thai. 2002 Feb;85(2):154-61. PMID 12081113
- [Result] Ayhan E, Kesmezacar H, Akgun I. Intraarticular injections (corticosteroid, hyaluronic acid, platelet rich plasma) for the knee osteoarthritis. World J Orthop. 2014 Jul 18;5(3):351-61. doi: 10.5312/wjo.v5.i3.351. eCollection 2014 Jul 18. PMID 25035839
- [Result] Huang Y, Liu X, Xu X, Liu J. Intra-articular injections of platelet-rich plasma, hyaluronic acid or corticosteroids for knee osteoarthritis : A prospective randomized controlled study. Orthopade. 2019 Mar;48(3):239-247. doi: 10.1007/s00132-018-03659-5. PMID 30623236
- [Result] Uslu Guvendi E, Askin A, Guvendi G, Kocyigit H. Comparison of Efficiency Between Corticosteroid and Platelet Rich Plasma Injection Therapies in Patients With Knee Osteoarthritis. Arch Rheumatol. 2017 Nov 2;33(3):273-281. doi: 10.5606/ArchRheumatol.2018.6608. eCollection 2018 Sep. PMID 30632533
- [Result] Dai WL, Zhou AG, Zhang H, Zhang J. Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis: A Meta-analysis of Randomized Controlled Trials. Arthroscopy. 2017 Mar;33(3):659-670.e1. doi: 10.1016/j.arthro.2016.09.024. Epub 2016 Dec 22. PMID 28012636
- [Result] Bennell KL, Hunter DJ, Paterson KL. Platelet-Rich Plasma for the Management of Hip and Knee Osteoarthritis. Curr Rheumatol Rep. 2017 May;19(5):24. doi: 10.1007/s11926-017-0652-x. PMID 28386761
- [Result] Parrish WR, Roides B. Physiology of blood components in wound healing: an appreciation of cellular co-operativity in platelet rich plasma action. J Exerc Sports Orthop 2017;4:1-14.
- [Result] Kabiri A, Esfandiari E, Esmaeili A, Hashemibeni B, Pourazar A, Mardani M. Platelet-rich plasma application in chondrogenesis. Adv Biomed Res. 2014 Jun 25;3:138. doi: 10.4103/2277-9175.135156. eCollection 2014. PMID 25161985
- [Result] Meheux CJ, McCulloch PC, Lintner DM, Varner KE, Harris JD. Efficacy of Intra-articular Platelet-Rich Plasma Injections in Knee Osteoarthritis: A Systematic Review. Arthroscopy. 2016 Mar;32(3):495-505. doi: 10.1016/j.arthro.2015.08.005. Epub 2015 Oct 1. PMID 26432430
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Amarase C, Tanavalee A, Veerasethsiri P, Ngarmukos S. Outcome measurements following total knee arthroplasty. JRCOST 2015;39:35-42.
- [Result] Riboh JC, Saltzman BM, Yanke AB, Fortier L, Cole BJ. Effect of Leukocyte Concentration on the Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis. Am J Sports Med. 2016 Mar;44(3):792-800. doi: 10.1177/0363546515580787. Epub 2015 Apr 29. PMID 25925602
- [Result] Abbas A, Du JT, Dhotar HS. The Effect of Leukocyte Concentration on Platelet-Rich Plasma Injections for Knee Osteoarthritis: A Network Meta-Analysis. J Bone Joint Surg Am. 2022 Mar 16;104(6):559-570. doi: 10.2106/JBJS.20.02258. PMID 34826301
- [Result] Di Martino A, Boffa A, Andriolo L, Romandini I, Altamura SA, Cenacchi A, Roverini V, Zaffagnini S, Filardo G. Leukocyte-Rich versus Leukocyte-Poor Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis: A Double-Blind Randomized Trial. Am J Sports Med. 2022 Mar;50(3):609-617. doi: 10.1177/03635465211064303. Epub 2022 Feb 1. PMID 35103547